CLINICAL TRIAL: NCT02239523
Title: Management Strategies by an Orthopedic Department to Improve the Evaluation and Treatment of Osteoporosis.
Brief Title: Effectiveness or Orthopedic Intervention in Osteoporosis Management After a Fracture of the Hip With Cost-Benefit Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201497CTIL
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2018-09

CONDITIONS: Osteoporotic Fracture
Keywords: Pathologic fracture; Insufficiency fracture; Secondary fracture; Fracture with bone fragility; Osteoporosis; Bone loss; Osteopenia; Metabolic Bone Disease; Fragility fracture
MeSH Terms: conditions — Osteoporotic Fractures; Fractures, Spontaneous; Fractures, Stress; Osteoporosis; Bone Diseases, Metabolic | interventions — Methods; Absorptiometry, Photon; Diphosphonates; Denosumab; Teriparatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letter Group (Active Comparator): Patients will be given discharge letter that includes recommendation to discuss further testing and treatment with their primary care physician.
  Interventions: Procedure: Letter Group
- Intervention Group (Experimental): Patients will be given a pamphlet about osteoporosis and importance of treatment, have a bone density test (DEXA) arranged, be given a specific medication recommendation and monthly followup phone calls.
  Interventions: Procedure: Intervention Group

INTERVENTIONS:
Procedure: Letter Group — At time of discharge from the hospital, patients will be sent home with a letter that includes standard recommendations for evaluation and treatment for osteoporosis. This will be asked to give the letter to their primary care physician.
  Arms: Letter Group
Procedure: Intervention Group — The orthopedic department will be responsible for arranging bone density testing (DEXA) and recommending specific medication after discharge. A research assistant will call monthly to encourage treatment.
  Other Names: Intervention; Dual-energy X-ray absorptiometry; Bone density scan; Bisphosphonate; Prolia; Denosumab; Forteo; Teriparatide
  Arms: Intervention Group

SUMMARY:
Patients who present with fragility fractures are consistently under-evaluated and under-treated for underlying osteoporosis. This point of care represents a lost opportunity to prevent future fractures. The medical field treats the fracture as if the fall is the problem, but bone quality is the real problem. Studies have consistently shown that the recommendations of the International Osteoporosis Foundation and World Health Organization are not being followed. Orthopedics treats the patients for their fractures and primary care physicians focus on general health but no one is taking responsibility for bone health. Strategies to convince primary care to assume care have not succeeded. On the other hand, strategies where orthopedics takes some responsibility have shown success. This prospective 2-arm study will evaluate the success of effort by an academic orthopedic department in osteoporosis evaluation and treatment. We hypothesize that with greater effort by the orthopedic department, the better the adherence to standards of care. A cost benefit analysis will be made in parallel.

DETAILED DESCRIPTION:
Patients who present to the orthopedic department in a level I trauma center will be prospectively randomized into one of two groups:

Letter Group: At time of discharge, patients will be sent home with a discharge letter that includes standard recommendations for evaluation and treatment. They will be asked to give the letter to their primary care physician.

Intervention Group: There will be 4 interventions. The patient will be given a short pamphlet with explaining osteoporosis and the importance of treatment. The orthopedic department will perform a bone density testing (DEXA). They will be given a letter with a specific medication recommendation based on a protocol determined by our endocrinology department. They will be asked to give both DEXA and medication recommendation to their primary care doctor to initiate treatment. Finally, a research assistant will contact the patient monthly to encourage them to start treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients over age 50 with fragility fracture defined as a fall from standing or walking position

Exclusion Criteria:

* Patients with metastatic cancer
* Known metabolic bone disease
* End-of-life care
* Inability to provide consent
* Known MRSA carriers
* Fractures of the trochanter alone, shaft or peri-prosthetic fractures

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with osteoporosis that are appropriately treated | Determination of proper treatment will be made at 4 months after the fracture.
  Treatment will be determined based on a pre-determined algorithm by our endocrinology department. This will be based on patient factors and results of DEXA is not part of the algorithm. All patients with a fragility fracture of the hip, regardless of DEXA results will be considered for treatment.

SECONDARY OUTCOMES:
Percentage of patients who undergo DEXA scan. | Evaluation will be made 4 months after the initial fracture event.
  Whether or not the patients received the medication

OTHER OUTCOMES:
Cost benefit analysis | Evaluation will be made at time of discharge and up to 4 months from the fracture event.
  Cost analysis will be made for each patient during the hospitalization and for 3 months after the fracture to capture complications related to the initial event.

CONTACTS AND LOCATIONS:
Overall Officials: Gershon Zinger, MD MS, Principal Investigator — Shaare Zedek Medical Center, Jerusalem Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Rozental TD, Makhni EC, Day CS, Bouxsein ML. Improving evaluation and treatment for osteoporosis following distal radial fractures. A prospective randomized intervention. J Bone Joint Surg Am. 2008 May;90(5):953-61. doi: 10.2106/JBJS.G.01121. PMID 18451385
- [Background] Edwards BJ, Koval K, Bunta AD, Genuario K, Hahr A, Andruszyn L, Williams M. Addressing secondary prevention of osteoporosis in fracture care: follow-up to "own the bone". J Bone Joint Surg Am. 2011 Aug 3;93(15):e87. doi: 10.2106/JBJS.I.00540. PMID 21915530
- [Background] Gardner MJ, Brophy RH, Demetrakopoulos D, Koob J, Hong R, Rana A, Lin JT, Lane JM. Interventions to improve osteoporosis treatment following hip fracture. A prospective, randomized trial. J Bone Joint Surg Am. 2005 Jan;87(1):3-7. doi: 10.2106/JBJS.D.02289. PMID 15634808
- [Derived] Zinger G, Sylvetsky N, Levy Y, Steinberg K, Bregman A, Yudkevich G, Peyser A. Early benefits of a secondary fracture prevention programme. Hip Int. 2023 Mar;33(2):332-337. doi: 10.1177/11207000211027476. Epub 2021 Jun 27. PMID 34180292